CLINICAL TRIAL: NCT03897452
Title: NeoFent-I Study; Fentanyl Treatment in Newborn Infants; a Pharmacokinetic, Pharmacodynamic and Pharmacogenetic Study. Prestudy to NeoOpioid; No Pain During Infancy by Adapting Off-patent Medicines. EU FP7:HEALTH - 2007-4.2-1
Brief Title: NeoFent-I Study; Fentanyl Treatment in Newborn Infants; a Pharmacokinetic, Pharmacodynamic and Pharmacogenetic Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Elisabeth Norman, MD, PhD, Senior Consultant, Lund University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU-Grant 223767; 2011-000310-19 (EudraCT Number)
Record Dates: First submitted 2019-02-13; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Pain
Keywords: analgesia; neonates; procedural pain; pain assessment; physiological response; pharmacogenetics
MeSH Terms: conditions — Pain; Agnosia; Pain, Procedural | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fentanyl for procedural pain (Experimental): A dose of Fentanyl 5 microgram/ml, 0.5 microgram/kg (anticipated medium pain) or 2 microgram/kg (anticipated strong pain) will be given prior to a painful procedure during NICU-care. Repeated doses or complementary analgesics will be administered according to pain assessment and clinical judgement.
  This is not an RCT with several arms.
  Interventions: Drug: Fentanyl (5 microgram/ml) prediluted ampoules

INTERVENTIONS:
Drug: Fentanyl (5 microgram/ml) prediluted ampoules — Bolus; Fentanyl (5 microgram/ml) 0,5 microgram/kg (0.1 ml/kg) is administered over 1 min starting 3-5 min before the lighter skin breaking procedure.
  Fentanyl (5 microgram/ml) 2 microgram/kg is administered over 10 min before the start of the more painful procedur ( pleura drainage or tracheal intubation).

SUMMARY:
The study will assess the efficacy of fentanyl using a pharmacokinetic/pharmacodynamic (PK/PD) model where the concentration of the drug is related to effect curve (pain score change in response to standardized procedural pain). Further cortical, physiological and biochemical responses to fentanyl will be assessed, elucidating the feasibility before the main study project (NeoOpioid) start.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for analgesia before any of following procedures;

  1. insertion of peripheral IV-catheter
  2. insertion of arterial cannula
  3. insertion of chest tube
  4. other skin breaking procedure.
* Possibility to obtain blood samle after the procedure (indwelling line)
* Infants all gestational ages.
* Postnatal age 0-28 days
* Informed written parental concent

Exclusion Criteria:

* Concurrent or previous opioid administration (72 h interval required)
* Abdominal surgery
* Major chromosomal anomaly
* Neonatal encephalopathy
* Use of muscle relaxant
* Hypothermia treatment after hypoxic-ischemic insult
* Clinical or biochemical evidence of hepatic failure
* Participation in other intervention trial

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics; fentanyl clearance | 48 hours
  Serum concentration will be analysed and the clearance will be calculated with NONMEM pharmacokinetics.
Pharmacokinetics; fentanyl clearance | 6 hours
  The serum concentration values will be analysed as Area under the curve, AUC
Pharmacodynamics; Amplitude integrated electroencephalography (aEEG) | 6 hours
  Background activity
Pharmacodynamics; Amplitude integrated electroencephalography (aEEG), | 6 hours
  Seizure activity

SECONDARY OUTCOMES:
Pharmacodynamics, change in vital parameters | 6 hours
  Change in heart rate
Pharmacodynamics, change in vital parameters | 6 hours
  Change in mean arterial blood pressure
Pharmacodynamics, change in vital parameters | 6 hours
  Change in near infrared spectroscopy
Pharmacodynamics, behavioural response | 6 hours
  Pain assessment with the Premature Infant Pain Profile-revised (PIPP) score for procedural pain (0-21, with the highest value if strong pain in extremely preterm infants)
Pharmacodynamics, hormonal response | 48 hours
  Blood levels of cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Vineta Fellman, Professor, Principal Investigator — Dep. of Pediatrics, Lund University, Sweden
Locations (1):
- Neonatal Intensive Care Unit, Skåne University Hospital, Lund, Sweden